CLINICAL TRIAL: NCT03969238
Title: Utilizing Helpline for Opioid Dependence Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Nassima Ait-Daoud Tiouririne, Associate Professor, Director of UVA Center for Leading Edge Addiction Research, University of Virginia
Other Study IDs: 21376
Record Dates: First submitted 2019-03-27; First posted 2019-05-31 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Opioid Dependence
Keywords: opioid dependence; pain management
MeSH Terms: conditions — Opioid-Related Disorders; Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients/Providers: Of the1,000 participants: (1) 900 will enroll as participants who use the helpline resources via verbal consent and (2) 100 will enroll as providers via online consent prior to survey data collection.
  Interventions: Behavioral: Helpline

INTERVENTIONS:
Behavioral: Helpline — This helpline will aim to provide patients with new diagnosis of pain who are prescribed opioids, access to education, support and free behavioral technique to help manage their pain such as mindfulness exercises. For those with opioid use disorder, the helpline will offer support in the form of education about the disorder, opioid withdrawal symptoms, risks of overdoses, and a variety of services such as help reach appropriate care with MAT licensed providers, information on FDA-approved MAT and naloxone, and, in some cases, behavioral intervention to keep patients engaged in treatment. The opioid helpline will provide a central resource for direct services and a portal for community services. It will also serve as a referral resource for health-care professionals.

SUMMARY:
The investigator propose to develop an opioid telephone helpline, where trained counselors and educators provide referral, educational and targeted interventions and support to individuals interested in addressing their addiction or needing help with managing their pain. The proposed application builds on "tobacco quit line" efforts, a nationally-adopted telephone-based service, providing education materials, access to cessation medication and counseling against tobacco use. Similar to tobacco quit line; the proposed telephone based services will remove barriers to treatment as they help individuals at the exact time of need. The helpline will also educate individuals with new onset pain about pain expectations, relaxation techniques, use of pharmacology and psychotherapy for treatment in addition to providing support for coping and reducing dependency on prescription opioids. It will be a low cost, easily accessible and utilizable technology to augment the clinical outcome of medication assisted treatment of opioid use disorder and pain management.

DETAILED DESCRIPTION:
The proposed specific aims are to:

1. Test if the helpline is a resourceful tool for patients with opioid use disorder looking for referrals and support to access treatment. The opioid helpline will provide individuals with opioid use disorder seeking treatment, direct access to a live person who can answer questions regarding referrals and various treatment programs. The helpline will also follow-up on treatment compliance and offer support and motivational techniques for these individuals to stay engaged in treatment
2. Test if the helpline is a resourceful tool for patients with new onset of pain or chronic pain being prescribed opioids. The opioid helpline will provide these individuals the necessary educational materials on managing pain safely while avoiding misuse. It will offer free imagery guided meditation and other non-pharmacological tools to help with pain management.
3. Test if providers find the opioid helpline helpful and resourceful for their practice and are willing to refer patients to the helpline.

ELIGIBILITY:
Inclusion Criteria:

Participant Criteria:

1. Age greater than or equal to 18 years.
2. A formal diagnosis of Opioid Use Disorder (OUD) by a health care provider or
3. If no formal diagnosis of OUD, having a self-reported concern with opioid use or addiction.
4. An individual seeking to reduce opioid use.
5. An individual concerned about opioids prescribed for management of new-onset pain or chronic pain.

Provider Criteria:

1. University of Virginia: Providers of any specialties within VA including dentists that prescribes opioids.
2. County of Wise: Providers of any specialties including dentists that prescribes opioids.

Exclusion Criteria:

Participant Criteria:

1. Individuals under 18 years of age.
2. Individuals seeking treatment for non-opioid substance use disorders
3. Individuals who have no pain issues
4. Individuals located outside of Virginia.

Provider Criteria:

Providers outside the designated regions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to pilot this model in a small rural area with low accessibility to specialized treatment. We will specifically target the area of county of Wise as it is an area with one of the highest rate of opioid addiction and overdose related deaths in the state.
  UVA hospital: we plan to pilot this model at UVA hospital because it is a health care system offering care to a diverse population from urban and rural areas.
  The providers will be educated regarding the goals and objectives of the helpline: Any specialty physicians, nurses including dentists that prescribes opioids within Virginia They will be asked to have flyers about the helpline in their office and refer patients who are prescribed opioids to get more support from the helpline.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Participant Opioid Helpline Survey | up to a year
  Primary outcomes measure the rating of the Helpline by the patients. They will be sent surveys that will ask the patients to rate the services they receive on a scale of 1 to 10, with 1 meaning they are very dissatisfied and 10 meaning they are very satisfied.
Provider Opioid Helpline Survey | up to a year
  Primary outcomes measure the rating of the Helpline by the providers. They will be sent surveys that will ask the providers to rate the services they receive on a scale of 1 to 10, with 1 meaning they are very dissatisfied and 10 meaning they are very satisfied.

SECONDARY OUTCOMES:
Number of participants reached versus called. | up to a year
  Total number of contacts to the Helpline compared to the number that prescreened and the number consented.
Number of participants who continued to access the services of Helpline | up to a year
  The investigator will measure the number of participants who continued to access the services of Helpline up to a year.
New General Self-Efficacy Measure | up to a year
  By using this survey, the investigator will determine the participant's ability to handle the situation that prompted the participant to call the Helpline originally.
Opioid Helpline Study Screen Form | up to a year
  This will be use to collect demographic information for individuals who self-identify as needing help or resources from the Helpline.
Referral follow-ups | up to a year
  Assess which referrals were followed up on by the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Nassima Ait-Daoud Tiouririne, M.D., Principal Investigator — University of Virginia
Locations (1):
- UVA Center for Leading Edge Addiction Research, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No